CLINICAL TRIAL: NCT00279994
Title: Exercise Therapy in Patients With Peripheral Arterial Disease: the Costs and Effectiveness of Physiotherapeutic Supervision With or Without Therapy Feedback Versus a "go Home and Walk" Advice
Brief Title: (Cost) Effectiveness Study of Exercise Therapy in Patients With Peripheral Arterial Disease
Acronym: EXITPAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Atrium Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Maastricht University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 945-06-252
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Intermittent Claudication
Keywords: Intermittent claudication; Exercise therapy; Therapy feedback; Accelerometer; Physiotherapy; PAD;; peripheral arterial disease according to Fontaine stage II)
MeSH Terms: conditions — Intermittent Claudication | interventions — Exercise Therapy

INTERVENTIONS:
Procedure: Exercise therapy
Device: Accelerometer (PAM; Personal Activity Monitor)
Procedure: Oral Exercise Therapy advise

SUMMARY:
The purpose of this study is to determine if supervised exercise therapy in a physiotherapeutic setting, with or without therapy feedback, is more (cost-)effective than exercise therapy based on a 'go home and walk' advice without supervision, for patients with PAD stage II (Fontaine).

DETAILED DESCRIPTION:
Exercise therapy (ET) is considered to be the main conservative treatment for patients with intermittent claudication (IC) and is documented to be effective, especially when supervised. However, wide scale introduction of supervised ET in the Netherlands would lead to a substantial increase of health care costs compared to current practice, while the cost-effectiveness of supervised ET is uncertain. ET follows a pattern of short walking periods that induce discomfort of moderate intensity and short rest periods. The psychological, metabolic, and mechanical alterations that occur during exercise stimulate an adaptive response that ultimately reduces the symptoms. The optimal therapy regimen depends to a large extent on home-based exercises, which require discipline from the patient. Currently, the main prescription for ET for patients with IC in the Netherlands is a single 'go home and walk' advice, without supervision or follow-up. There is no evidence to support the effectiveness of this advice and compliance is low. In studies comparing the 'go home and walk' advice to supervised ET, a large advantage for supervised ET was present. The inadequate use of the main conservative treatment for peripheral arterial disease (PAD) contributes to a gradual progression of this condition, a decrease in quality of life, and an increasing number of vascular interventions. Furthermore, with adequate ET, hypertension, hypercholesterolemia, overweight, and diabetes, if present, is better regulated.

ELIGIBILITY:
Inclusion Criteria:

* PAD stage II
* Ankle-brachial index below 0.9
* Maximal walking distance of 500 meters or less

Exclusion Criteria:

* prior ET
* previous peripheral vascular interventions
* no insurance for physiotherapy
* insufficient command of the Dutch language
* serious cardiopulmonary limitations (NYHA-3-4)
* previous amputation
* psychiatric instability
* other serious co-morbidity prohibiting physical training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-12; Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
maximal walking distance

SECONDARY OUTCOMES:
pain-free walking distance
blood pressure
fasting glucose
fasting cholesterol
lipids profile
body weight
co-morbidity
vascular interventions
mortality
medical and non-medical costs
compliance
quality of life
impairment
complaints

CONTACTS AND LOCATIONS:
Overall Officials: Joep A.W. Teijink, PhD MD, Principal Investigator — Atrium Medical Centre Parkstad; Martin H. Prins, Prof. PhD MD, Study Chair — Maastricht University
Locations (1):
- Atrium Medical Centre, Heerlen, P.O.box 4446, Netherlands

REFERENCES:
- [Background] Stewart KJ, Hiatt WR, Regensteiner JG, Hirsch AT. Exercise training for claudication. N Engl J Med. 2002 Dec 12;347(24):1941-51. doi: 10.1056/NEJMra021135. No abstract available. PMID 12477945
- [Background] Patterson RB, Pinto B, Marcus B, Colucci A, Braun T, Roberts M. Value of a supervised exercise program for the therapy of arterial claudication. J Vasc Surg. 1997 Feb;25(2):312-8; discussion 318-9. doi: 10.1016/s0741-5214(97)70352-5. PMID 9052565
- [Background] Savage P, Ricci MA, Lynn M, Gardner A, Knight S, Brochu M, Ades P. Effects of home versus supervised exercise for patients with intermittent claudication. J Cardiopulm Rehabil. 2001 May-Jun;21(3):152-7. doi: 10.1097/00008483-200105000-00006. PMID 11409225
- [Background] Regensteiner JG, Meyer TJ, Krupski WC, Cranford LS, Hiatt WR. Hospital vs home-based exercise rehabilitation for patients with peripheral arterial occlusive disease. Angiology. 1997 Apr;48(4):291-300. doi: 10.1177/000331979704800402. PMID 9112877
- [Background] Cheetham DR, Burgess L, Ellis M, Williams A, Greenhalgh RM, Davies AH. Does supervised exercise offer adjuvant benefit over exercise advice alone for the treatment of intermittent claudication? A randomised trial. Eur J Vasc Endovasc Surg. 2004 Jan;27(1):17-23. doi: 10.1016/j.ejvs.2003.09.012. PMID 14652832
- [Background] Degischer S, Labs KH, Hochstrasser J, Aschwanden M, Tschoepl M, Jaeger KA. Physical training for intermittent claudication: a comparison of structured rehabilitation versus home-based training. Vasc Med. 2002 May;7(2):109-15. doi: 10.1191/1358863x02vm432oa. PMID 12402991
- [Background] Brandsma JW, Robeer BG, van den Heuvel S, Smit B, Wittens CH, Oostendorp RA. The effect of exercises on walking distance of patients with intermittent claudication: a study of randomized clinical trials. Phys Ther. 1998 Mar;78(3):278-86; discussion 286-8. doi: 10.1093/ptj/78.3.278. PMID 9520973
- [Background] Gardner AW, Poehlman ET. Exercise rehabilitation programs for the treatment of claudication pain. A meta-analysis. JAMA. 1995 Sep 27;274(12):975-80. PMID 7674529
- [Background] Leng GC, Fowler B, Ernst E. Exercise for intermittent claudication. Cochrane Database Syst Rev. 2000;(2):CD000990. doi: 10.1002/14651858.CD000990. PMID 10796572
- [Background] Bartelink ML, Stoffers HE, Biesheuvel CJ, Hoes AW. Walking exercise in patients with intermittent claudication. Experience in routine clinical practice. Br J Gen Pract. 2004 Mar;54(500):196-200. PMID 15006125
- [Background] Dormandy J, Heeck L, Vig S. The natural history of claudication: risk to life and limb. Semin Vasc Surg. 1999 Jun;12(2):123-37. PMID 10777239
- [Background] Hooi JD, Kester AD, Stoffers HE, Overdijk MM, van Ree JW, Knottnerus JA. Incidence of and risk factors for asymptomatic peripheral arterial occlusive disease: a longitudinal study. Am J Epidemiol. 2001 Apr 1;153(7):666-72. doi: 10.1093/aje/153.7.666. PMID 11282794
- [Background] Willigendael EM, Teijink JA, Bartelink ML, Boiten J, Moll FL, Buller HR, Prins MH. Peripheral arterial disease: public and patient awareness in The Netherlands. Eur J Vasc Endovasc Surg. 2004 Jun;27(6):622-8. doi: 10.1016/j.ejvs.2004.02.019. PMID 15121113
- [Background] Gardner AW, Katzel LI, Sorkin JD, Bradham DD, Hochberg MC, Flinn WR, Goldberg AP. Exercise rehabilitation improves functional outcomes and peripheral circulation in patients with intermittent claudication: a randomized controlled trial. J Am Geriatr Soc. 2001 Jun;49(6):755-62. doi: 10.1046/j.1532-5415.2001.49152.x. PMID 11454114
- [Background] McDermott MM, Liu K, O'Brien E, Guralnik JM, Criqui MH, Martin GJ, Greenland P. Measuring physical activity in peripheral arterial disease: a comparison of two physical activity questionnaires with an accelerometer. Angiology. 2000 Feb;51(2):91-100. doi: 10.1177/000331970005100201. PMID 10701716
- [Background] Sieminski DJ, Gardner AW. The relationship between free-living daily physical activity and the severity of peripheral arterial occlusive disease. Vasc Med. 1997 Nov;2(4):286-91. doi: 10.1177/1358863X9700200402. PMID 9575600
- [Background] Sieminski DJ, Cowell LL, Montgomery PS, Pillai SB, Gardner AW. Physical activity monitoring in patients with peripheral arterial occlusive disease. J Cardiopulm Rehabil. 1997 Jan-Feb;17(1):43-7. doi: 10.1097/00008483-199701000-00006. PMID 9041070
- [Background] Moreland JD, Thomson MA, Fuoco AR. Electromyographic biofeedback to improve lower extremity function after stroke: a meta-analysis. Arch Phys Med Rehabil. 1998 Feb;79(2):134-40. doi: 10.1016/s0003-9993(98)90289-1. PMID 9473993
- [Background] Weatherall M. Biofeedback or pelvic floor muscle exercises for female genuine stress incontinence: a meta-analysis of trials identified in a systematic review. BJU Int. 1999 Jun;83(9):1015-6. doi: 10.1046/j.1464-410x.1999.00091.x. PMID 10368247
- [Background] Beddy P, Neary P, Eguare EI, McCollum R, Crosbie J, Conlon KC, Keane FB. Electromyographic biofeedback can improve subjective and objective measures of fecal incontinence in the short term. J Gastrointest Surg. 2004 Jan;8(1):64-72; discussion 71-2. doi: 10.1016/j.gassur.2003.10.005. PMID 14746837
- [Background] Dolan P, Gudex C, Kind P, Williams A. A social tariff for EuroQol: results from a UK general population survey. York Centre for Health Economics Discussion Paper 1381990 University of York, 1995
- [Background] Nielsen SL, Larsen B, Prahl M, Jensen CT, Jensen BE, Wenkens V. [Hospital training compared with home training in patients with intermittent claudication]. Ugeskr Laeger. 1977 Nov 14;139(46):2733-6. No abstract available. Danish. PMID 595156
- [Background] Nielsen SL, Gyntelberg F, Larsen B, Lassen NA. Hospital versus home training, a clinical trial. Aktuelle probleme in der angiology 1975;30:121-126
- [Background] Ambrosetti M, Salerno M, Boni S, Daniele G, Tramarin R, Pedretti RF. Economic evaluation of a short-course intensive rehabilitation program in patients with intermittent claudication. Int Angiol. 2004 Jun;23(2):108-13. PMID 15507886
- [Background] de Vries SO, Visser K, de Vries JA, Wong JB, Donaldson MC, Hunink MG. Intermittent claudication: cost-effectiveness of revascularization versus exercise therapy. Radiology. 2002 Jan;222(1):25-36. doi: 10.1148/radiol.2221001743. PMID 11756701
- [Background] Treesak C, Kasemsup V, Treat-Jacobson D, Nyman JA, Hirsch AT. Cost-effectiveness of exercise training to improve claudication symptoms in patients with peripheral arterial disease. Vasc Med. 2004 Nov;9(4):279-85. doi: 10.1191/1358863x04vm570oa. PMID 15678620
- [Derived] Gommans LN, Scheltinga MR, van Sambeek MR, Maas AH, Bendermacher BL, Teijink JA. Gender differences following supervised exercise therapy in patients with intermittent claudication. J Vasc Surg. 2015 Sep;62(3):681-8. doi: 10.1016/j.jvs.2015.03.076. PMID 26304482
- [Derived] Nicolai SP, Hendriks EJ, Prins MH, Teijink JA; EXITPAD study group. Optimizing supervised exercise therapy for patients with intermittent claudication. J Vasc Surg. 2010 Nov;52(5):1226-33. doi: 10.1016/j.jvs.2010.06.106. Epub 2010 Aug 8. PMID 20692797